CLINICAL TRIAL: NCT05443932
Title: Dapagliflozin and Hydrochlorothiazide Treatment in Recurring Kidney Stone Patients - a Randomised Single Center Cross-over Study
Brief Title: Dapagliflozin and Hydrochlorothiazide in Recurring Kidney Stone Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Zeljko Kikic, Assoc.Prof.Priv.Doz.Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Urolithiasis
Record Dates: First submitted 2022-03-15; First posted 2022-07-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Urolithiasis; Hyperoxaluria
Keywords: Urolithiasis; Hyperoxaluria
MeSH Terms: conditions — Urolithiasis; Hyperoxaluria | interventions — dapagliflozin; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: There won´t be comparator arms in our study. Instead, the investigators plan to do blood- and 24h-urine screenings including oxalate and citrate as well as metabolomics tests out of blood and urine samples at crucial points of time of the study to get baseline and therapeutic data of the participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Washout Phase and treatment arms (Other): At first there will be wash-out phase I with daily placebo administration for all participants. All patients will receive blood- and 24h-urine screenings in week 0 and 6 to get baseline data and also a low-dose native CT of the urinary tract in week 6. In preparation of the HCT phase all participants will daily receive an oral placebo.
  In week 7 the HCT phase will start and all patients will receive an oral therapy with 50mg of HCT daily; the treatment response will be evaluated by blood- and urine test after 4 weeks of therapy (week 10).
  After that, in washout phase II, the same test as before will be performed in week 0 and 6 (weeks 15 and 20).
  At the end another therapy phase with an oral administration of 10mg dapagliflozin daily will be performed; the treatment response will be evaluated by blood- and urine test after 4 weeks of therapy (week 25).
  Finally, the same tests as before will be performed in wash-out phase III in week 0 and 6 (weeks 29 and 34).
  Interventions: Drug: Dapagliflozin; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Dapagliflozin — 10mg Dapagliflozin daily for 8 weeks
Drug: Hydrochlorothiazide — 50mg Hydrochlorothiazide daily for 8 weeks

SUMMARY:
Current prevention strategies in patients with recurrence of kidney stones show especially in high-risk patients a diversely and in the long-term not successful outcome in a sustainable number of cases. Recent studies have revealed that Dapagliflozin has the potential to decrease risk and incidence of urolithiasis events especially in patients suffering from Diabetes. The investigators propose that Dapagliflozin has the potential to increase the metabolic situation of hyperoxaluric patients with recurrence of urolithiasis. The investigators therefore test whether Dapagliflozin can decrease the oxalate excretion compared to the current strategy with Hydrochlorothiazide. The study may open up a new way of preventing urolithiasis in patients with high-risk of recurring urolithiasis.

ELIGIBILITY:
Inclusion Criteria:

• Calcium-oxalate stone formers with high risk of reoccurrence defined as:

* At least two symptomatic or surgically treated kidney stones within the last 10 years and/or
* Single stone kidney formers with risk factors including: a.) Positive medical family history on kidney stone formations of at least one blood related relative in the first degree or at least two blood related relatives in the second degree and/ or b.) Onset of kidney stone formations within the third life decade or earlier and/ or c.) Metabolic syndrome d.) Obesity (BMI ≥ 30 kg/m²)

Exclusion Criteria:

* Age < 18 years
* Malabsorption disorder
* eGFR < 30 ml/min/1,73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Δ of urinary oxalate excretion | 8 weeks
  As the primary endpoint the investigators defined the change of the urine oxalate excretion assessed by 24 h hour urine by 25% after 8 weeks of SGLT-2 inhibitor therapy compared to the baseline value that was collected in the washout phase before the treatment period. (Δ week0 and week 8 in mmol/L)

SECONDARY OUTCOMES:
Δ of urinary calcium excretion | 8 weeks
  Reduction of the urine calcium excretion assessed by 24 h hour urine by 25% after 8 weeks of SGLT-2 inhibitor therapy compared to the baseline value that was collected in the washout phase before the treatment period. (Δ week0 and week 8 in mmol/L)
Change of serum kreatinine | 8 weeks
  Change of serum kreatinine (in mg/dL) assessed by blood collection after 8 weeks of SGLT-2 inhibitor therapy compared to the baseline value that was collected in the washout phase before the treatment period.
Frequency of urolithiasis | 12 months
  Frequency of sympothomatic or treatment worthy urolithiasis events within the 12 month lasting afterward study period. (in events/ person/ year)
Tolerability of SGLT-2inhibitor therapy | 8 weeks
  Tolerability of the SGLT-2 inhibitors within 8 weeks lasting therapy phase assessed by a physician in [Type of adverse event; Start (date and time); End (date and time); Severity (mild, moderate, severe); Serious (no / yes); Unexpected (no / yes); Outcome (resolved, resolving, not resolved, resolved with sequelae, unknown, fatal); Relation to study drug (Related/ Probably/ Possibly/ Unlikely/ Not related/ Not assessable)].
Change of eGFR | 8 weeks
  Change of eGFR (in ml/min/1,73 m2) that was calculated from serum kreatinine that was assessed by blood collection after 8 weeks of SGLT-2 inhibitor therapy compared to the baseline value that was collected in the washout phase before the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria